CLINICAL TRIAL: NCT04549363
Title: Characterization of Corneal Epithelial Changes in Participants Treated With Belantamab Mafodotin (GSK2857916)
Brief Title: Characterization of Corneal Epithelial Changes in Participants Treated With Belantamab Mafodotin
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study has been terminated for reasons pertaining to feasibility
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 214098
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Results first posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Multiple Myeloma
Keywords: Belantamab mafodotin; Impression cytology; Superficial keratectomy; Relapsed/Refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants undergoing IC (Experimental): IC will be performed on some participants who received or are receiving treatment with belantamab mafodotin for RRMM and have objective evidence of keratopathy with corneal deposits on slit-lamp and/or confocal microscopy examination and who do not agree to undergo SK.
  Interventions: Drug: Belantamab mafodotin
- Participants undergoing SK (Experimental): SK will be performed on some participants who received or are receiving treatment with belantamab mafodotin for RRMM and have objective evidence of keratopathy with corneal deposits on slit-lamp and/or confocal microscopy examination.
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin is a first-in-class immunoconjugate that targets B cell maturation antigen (BCMA), which is highly expressed on malignant plasma cells.

SUMMARY:
This study will be available to any participant who has received or is currently receiving belantamab mafodotin treatment through either a clinical trial, an access program, or a physician prescription. Participants do not need to be on active treatment. The purpose of this study is to gain a more complete understanding of the pathophysiology of the corneal events seen in some participants with relapsed/refractory multiple myeloma (RRMM) treated with belantamab mafodotin. A superficial corneal epithelial tissue specimen will be obtained by performing impression cytology (IC) or superficial keratectomy (SK) procedure in participants treated with belantamab mafodotin. The procedure will only be performed in one eye, most affected by the corneal epithelial changes. This specimen will undergo pathologic examination and composition analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 years or older (at the time consent is obtained).
* Capable of providing signed written informed consent, which includes compliance with the requirements and restrictions listed on the consent form.
* Participants with RRMM who have received or are currently receiving treatment with belantamab mafodotin and diagnosed with microcyst-like epithelial changes (MECs) on slit-lamp examination or confocal microscopy, with or without symptoms, in at least one eye.

  a) If participants only had superficial punctate keratopathy with no evidence of MEC's they are not eligible.
* If undergoing SK procedure, treating provider has determined there is no excessive risk to the participant.

Exclusion Criteria:

* Any serious and or/unstable medical or psychiatric disorder, or other conditions that could interfere with the participant's safety.
* Any excess risk of delayed wound healing (For example, diabetes mellitus).
* Do not meet criteria specified by the study or program through which they would receive belantamab mafodotin.
* Any participant taking concurrent medication that may affect the cornea (that is. amiodarone, some chloroquines).
* Any participant with decreased corneal sensation.
* Eye infections, including infectious keratopathy, stye, blepharitis, and conjunctivitis.
* An active uveitis including anterior, posterior, or panuveitis in either eye.
* Permanent legal blindness in the fellow (non-study) eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2022-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- United States (6):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Westwood, Kansas
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Lee V, Hultcrantz M, Petrone S, Lewis EW, Banna H, Lichtman E, Thulasi P, Quick AA, Jeng BH, Sunshine SB, Francis JH, Canestraro J, Farooq AV, Clements P, Robertson N, Burman M, McKevitt T, Struemper H, Weir L. Characterization of Belantamab Mafodotin-Induced Corneal Changes in Patients With Multiple Myeloma. JAMA Ophthalmol. 2025 Jun 1;143(6):507-514. doi: 10.1001/jamaophthalmol.2025.1008. PMID 40338596

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has been terminated for reasons pertaining to feasibility.
Pre-assignment Details: Out of the 16 participants enrolled, 7 were screen failures, 9 participants were allocated to undergo Impression Cytology (IC)/ Superficial Keratectomy (SK) procedure.
Groups:
- Participants Allocated to Undergo Impression Cytology Procedure: A superficial corneal epithelial tissue specimen was obtained by performing impression cytology (IC) procedure in participants with relapsed/refractory multiple myeloma (RRMM) treated with belantamab mafodotin. The procedure was only performed in one eye. Participants did not need to be on active treatment.
- Participants Allocated to Undergo Superficial Keratectomy Procedure: A superficial corneal epithelial tissue specimen was obtained by performing superficial keratectomy (SK) procedure in participants with relapsed/refractory multiple myeloma (RRMM) treated with belantamab mafodotin. The procedure was only performed in one eye. Participants did not need to be on active treatment.
Period: Overall Study
Arm/Group | Participants Allocated to Undergo Impression Cytology Procedure | Participants Allocated to Undergo Superficial Keratectomy Procedure
Started (All treated population) | 6 | 3
ICSK Population (IC or SK (ICSK) population is defined as participants from all-treated population who had a tissue sample collected using Impression Cytology (IC) or Superficial Keratectomy (SK) procedure, whether or not the specimen is evaluable.) | 6 | 3
EICSK Population (Evaluable IC or SK (EICSK) population included participants from all-treated population who had an evaluable tissue sample collected using IC or SK procedure. A tissue sample specimen were determined to be evaluable by the pathologist in the pathology report.) | 4 | 2
Completed | 6 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants Allocated to Undergo Impression Cytology Procedure | Participants Allocated to Undergo Superficial Keratectomy Procedure | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.5 (9.05) | 71.3 (8.50) | 69.4 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 0 | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Not Hispanic or Latino | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Abnormality in Composition of Corneal Epithelium After Administration of Belantamab Mafodotin
Description: Corneal tissue samples were collected to evaluate the composition of microcyst-like epithelium observed in participants treated with belantamab mafodotin.
Time Frame: Up to approximately 23 months
Population: EICSK population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Allocated to Undergo Impression Cytology Procedure | Participants Allocated to Undergo Superficial Keratectomy Procedure
Number analyzed (Participants) | 4 | 2
Participants | 4 | 2

2. Primary Outcome: Number of Participants With Abnormality in Pathologic Characteristics After Administration of Belantamab Mafodotin
Description: Corneal tissue samples were collected to evaluate pathologic characteristics observed in participants treated with belantamab mafodotin.
Time Frame: Up to approximately 23 months
Population: EICSK population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Allocated to Undergo Impression Cytology Procedure | Participants Allocated to Undergo Superficial Keratectomy Procedure
Number analyzed (Participants) | 4 | 2
Participants | 4 | 2

3. Secondary Outcome: Number of Participants With Imaging Data Showing Histopathologic Findings
Description: The eye was visualized using a slit-lamp microscope in a procedure room.
Time Frame: Up to approximately 23 months
Population: ICSK Population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Allocated to Undergo Impression Cytology Procedure | Participants Allocated to Undergo Superficial Keratectomy Procedure
Number analyzed (Participants) | 6 | 3
Participants | 2 | 3

4. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to approximately 23 months
Population: ICSK population
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Allocated to Undergo Impression Cytology Procedure | Participants Allocated to Undergo Superficial Keratectomy Procedure
Number analyzed (Participants) | 6 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse events (non-SAEs) and serious adverse events (SAEs) were collected up to approximately 23 months.
Description: Impression cytology or superficial keratectomy procedure (ICSK) population included participants from all-treated population who had a tissue sample collected using IC or SK procedure, whether or not the specimen is evaluable.
Arm/Group | Participants Allocated to Undergo Impression Cytology Procedure | Participants Allocated to Undergo Superficial Keratectomy Procedure
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/63/NCT04549363/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT04549363/SAP_001.pdf